CLINICAL TRIAL: NCT06582524
Title: A Phase 3 Open-Label Study of Safety, Pharmacokinetics, and Activity of Weekly Subcutaneous Pegzilarginase in Subjects <24 Months Old With Arginase 1 Deficiency
Brief Title: Pegzilarginase in Subjects <24 Months Old With Arginase 1 Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Immedica Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAEB1102-301A (Europe)
Record Dates: First submitted 2024-08-20; First posted 2024-09-03 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Arginase 1 Deficiency
MeSH Terms: conditions — Hyperargininemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weekly subcutaneous (SC) administration of pegzilarginase (Experimental): All subjects will receive a once weekly (QW) SC dose of pegzilarginase for 12 weeks
  Interventions: Drug: Pegzilarginase

INTERVENTIONS:
Drug: Pegzilarginase — SC administration of pegzilarginase over 12 weeks in subjects with ARG1-D who are < 24 months of age
  Other Names: Loargys

SUMMARY:
This is an open-label, multicentre study to evaluate the safety, PK, and activity (PD) of weekly subcutaneous (SC) administration of pegzilarginase in subjects with ARG1-D who are < 24 months of age. The study consists of a screening period of up to 4 weeks, a subsequent 12-week treatment period, and a safety follow-up period of 8 weeks.

DETAILED DESCRIPTION:
CAEB1102-301A is an open-label, single-arm, non-controlled, repeat dosing, multicentre study to evaluate the safety, PK, and activity (PD) of weekly SC administration of pegzilarginase over 12 weeks in subjects with ARG1-D who are < 24 months of age.

This study will consist of:

* A screening period of up to 4 weeks to ensure the subjects meet the study eligibility criteria and establish baseline plasma arginine
* A treatment period of 12 weeks
* A safety follow-up period of 8 weeks with visits 1 week and 8 weeks after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be < 24 months of age on the date of informed consent
2. Confirmed diagnosis of ARG1-D documented in medical records by at least 1 of the following methods:

   1. elevated plasma arginine levels
   2. a mutation analysis revealing a pathogenic variant
   3. red blood cell (RBC) arginase activity
3. Subjects must weigh > 8 kg due to clinical trial related blood collection volumes required
4. Written informed consent by parent/legal guardian, in accordance with national stipulations, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol
5. At least one value of plasma arginine ≥ 180 μM during screening
6. Documented confirmation from the Investigator and/or dietitian that the subject can:

   1. attempt to maintain a stable, age-appropriate level of protein consumption, including natural protein, and EAA supplementation within approximately ± 15% of dietitian recommended diet
   2. attempt to maintain current use of ammonia scavengers, if prescribed

Exclusion Criteria:

1. Other medical condition(s) or comorbidity(ies) that, in the opinion of the Investigator, would interfere with study compliance or data interpretation
2. Hyperammonaemic episode (plasma ammonia levels > 100 μM) with ≥ 1 symptom related to hyperammonaemia requiring hospitalisation or emergency room management within the 4 weeks before the first dose of study drug
3. Active infection requiring anti-infective therapy within < 2 weeks before first dose of study drug
4. Known active infection with human immunodeficiency virus, hepatitis B, or hepatitis C
5. History of hypersensitivity to polyethylene glycol (PEG) or any of the excipients included in the study drug that, in the judgment of the Investigator, puts the subject at unacceptable risk for AEs
6. Currently participating in another therapeutic clinical study or has received any investigational agent within 30 days (or 5 half-lives, whichever is longer) prior to first dose of study drug
7. Previous liver or haematopoietic stem cell transplant
8. Use of botulinum toxin within 16 weeks prior to first dose

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of pegzilarginase | From baseline up to 12 weeks
  To evaluate the effect of pegzilarginase on plasma arginine concentrations in subjects <24 months of age with arginase 1 deficiency (ARG1-D)

SECONDARY OUTCOMES:
To evaluate the safety of pegzilarginase | From baseline up to 12 weeks
  Safety assessments will include: adverse events (AEs), including hypersensitivity reactions (HSRs), injection site reactions (ISRs), safety labs and hyperammonaemic events
To characterize the pharmacokinetic (PK) profile of pegzilarginase | From baseline up to 12 weeks
  PK parameters with evaluation of half-life (T½)
To characterize the pharmacokinetic (PK) profile of pegzilarginase | From baseline up to 12 weeks
  PK parameters with evaluation on time to maximum observed concentration (Tmax)
To characterize the pharmacokinetic (PK) profile of pegzilarginase | From baseline up to 12 weeks
  PK parameters with evaluation of maximum observed concentration (Cmax)
To characterize the pharmacokinetic (PK) profile of pegzilarginase | From baseline up to 12 weeks
  PK parameters with evaluation on area under the plasma drug concentration-time curve
To evaluate the pharmacodynamic (PD) response of pegzilarginase | From baseline up to 12 weeks
  PD response evaluation including anti-drug antibodies (ADAs), levels of plasma arginine and ornithine
To describe changes in physical function | From baseline up to 12 weeks
  Changes in physical function after 12 weeks of pegzilarginase treatment as measured by Gross Motor Function Measure (GMFM)-66 Parts A through E, as age appropriate and feasible
To evaluate the safety of pegzilarginase | From baseline up to 12 weeks
  Safety assessments will include electrocardiograms (ECGs) to evalute P Wave, QRS Complex, QT Interval

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Rudebeck, PhD MSc BMedSc, Study Director — Immedica Pharma AB
Locations (3):
- Univ. Klinik für Kinder- und Jugendheilkunde Medizinische Universität, Graz, Austria
- Unidade de Doenças Metabólicas Pediatria, Hospital Santa Maria, Lisbon, Portugal
- Bradford Royal Infirmary Duckworth Lane, Bradford, United Kingdom

IPD SHARING:
Plan to Share IPD: No